CLINICAL TRIAL: NCT00050336
Title: A Phase 3 Randomized Study of Lonafarnib in Combination With Paclitaxel and Carboplatin vs. Placebo in Combination With Paclitaxel and Carboplatin in Patients With Non-Small Cell Lung Cancer
Brief Title: Study of Lonafarnib in Combination With Paclitaxel and Carboplatin in Patients With Non-Small Cell Lung Cancer (Study P01901)(TERMINATED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P01901
Record Dates: First submitted 2002-12-04; First posted 2002-12-05 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Carcinoma, Non-small-cell Lung; Metastases, Neoplasm
Keywords: Stage 3b or 4 (metastatic) non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — lonafarnib

INTERVENTIONS:
Drug: Lonafarnib (SARASAR)

SUMMARY:
The purpose of this study is to determine the overall survival of patients diagnosed with Stage 3b or 4 non-small cell lung cancer (NSCLC) treated with an oral Farnesyl Protein Transferase Inhibitor (Lonafarnib/SCH 66336) in combination with paclitaxel and carboplatin with that of patients treated with placebo in combination with paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Histologically or cytologically 3b or 4 (metastatic) non-small cell lung cancer. Patients must meet any subcriteria as detailed in the protocol.
* Age greater than or equal to 18 years old
* ECOG performance status of 0 to 1
* Prior diagnosis of brain metastases from NSCLC eligible provided that the brain metastases have been adequately treated, patient is neurologically stable and no new or progressive brain metastases identified.
* Meets protocol requirements for specified laboratory values
* Written informed consent
* Appropriate use of effective contraception if of childbearing potential
* Prior basal cell carcinoma or carcinoma in-situ of the cervix are eligible provided they have been treated with no evidence of disease

Exclusion Criteria:

* Prior chemotherapy for any stage of NSCLC
* Prior surgery or radiation therapy within the last 2 weeks or incomplete recovery from prior procedures or therapy
* Concurrent treatment or treatment within the last 2 years for any other malignancy
* Grade 2 or greater nausea or Grade 1 or greater vomiting (despite antiemetic medication)
* Medical conditions that would interfere with taking oral medications
* Patients with bone metastases as the only site of disease
* Pregnant or nursing women
* Known HIV positivity or AIDS-related illness
* Patients with significant QTc prolongation at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2002-12; Primary Completion 2004-02 (Actual); Study Completion 2004-03 (Actual)